CLINICAL TRIAL: NCT01496703
Title: Reasons for Dose Reduction of Mycophenolate Mofetil During the First Post-transplant Year in Renal Transplant Recipients and Its Impact on Graft Outcome: a Single-center Retrospective Analysis
Brief Title: Reasons for Mycophenolate Mofetil Dose Reduction and Impact on Graft Outcome in Renal Transplant Recipients
Status: Completed | Type: Observational
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Principal Investigator, Bert Bammens, Clinical Professor, Principal Investigator, Universitaire Ziekenhuizen KU Leuven
Other Study IDs: MMFreductionLeuven
Record Dates: First submitted 2011-12-17; First posted 2011-12-21 (Estimated); Last update posted 2011-12-21 (Estimated); Status verified 2011-12

CONDITIONS: Acute Rejection of Renal Transplant; Renal Graft Loss
Keywords: reasons for MMF dose reduction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- renal transplantation with MMF from day 1
  Interventions: Other: no intervention, this is an observational retrospective trial

INTERVENTIONS:
Other: no intervention, this is an observational retrospective trial — no intervention, this is an observational retrospective trial

SUMMARY:
Mycophenolate mofetil (MMF) decreases the risk of acute rejection and is associated with improved graft survival in renal transplant recipients. However, MMF-related side effects often necessitate dose reduction which may expose transplant recipients to a higher risk of acute rejection and graft loss. This study's aim was to examine the reasons for MMF dose reduction during the first year after kidney transplantation and its impact on acute rejection, overall and death-censored graft loss. Methods: Retrospective electronic file based analysis of all patients who underwent a single kidney transplantation in our center between 1996 and 2007 and were treated with MMF as part of their initial maintenance immunosuppressive protocol (n=749).

ELIGIBILITY:
Inclusion Criteria:

* All patients who received a single renal transplant at the University Hospitals of Leuven between April 1996 (when MMF was introduced in the Leuven renal transplant program) and February 2007 and were treated with MMF (Cellcept®, Roche) as part of their initial maintenance immunosuppressive regimen were included in this retrospective analysis.

Exclusion Criteria:

* If a patient underwent more than one kidney transplantation in the abovementioned 11-year period, only the last was considered.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients who received a single renal transplant at the University Hospitals of Leuven between April 1996 (when MMF was introduced in the Leuven renal transplant program) and February 2007 and were treated with MMF (Cellcept®, Roche) as part of their initial maintenance immunosuppressive regimen were included in this retrospective analysis. If a patient underwent more than one kidney transplantation in the abovementioned 11-year period, only the last was considered. No other exclusion criteria were applied.
Sampling Method: Non-Probability Sample
Enrollment: 749 (Actual)
Dates: Start 1996-01; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
reasons for dose reduction of MMF | 400 days post-transplantation

SECONDARY OUTCOMES:
occurence of acute rejection | 400 days post-transplantation
graft survival | 400 days post-transplantation

CONTACTS AND LOCATIONS:
Overall Officials: Bert Bammens, MD,PhD, Principal Investigator — Universitaire Ziekenhuizen KU Leuven
Locations (1):
- Universitaire Ziekenhuizen Leuven, Leuven, Belgium